CLINICAL TRIAL: NCT03587025
Title: Preemptive Analgesia With Amitryptyline for Prevention of Post-operative Pain in Women After Total Abdominal Hysterectomy: a Randomized Clinical Trial
Brief Title: Preemptive Analgesia With Amitryptyline for Prevention of Pain in Women After Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Antonio Henriques de França Neto, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMIP
Record Dates: First submitted 2015-07-08; First posted 2018-07-16 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative
Keywords: amitryptyline; Analgesia; Hysterectomy; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amitryptyline (Active Comparator): Patients who will be take amitryptyline, 75mg, only use, 30min before surgery.
  Interventions: Drug: Amitriptyline
- Placebo (Placebo Comparator): Patients who will be take placebo 30min before surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline compared with placebo for preemptive analgesia in women after abdominal hysterectomy.
  Arms: Amitryptyline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether amitryptyline is effective in the prevention of pain in women after a total abdominal hysterectomy.

DETAILED DESCRIPTION:
It will be performed a randomized clinical trial, double-blind, placebo-controlled, with two branches: one group receiving preemptive analgesia with amitryptyline and one receiving placebo. Blind procedures (blinding):

1. The participant does not know which group participates;
2. The evaluator does not know to which group it belongs to every individual;
3. The tablets provided to patients will be identical.

Study population All patients with total abdominal hysterectomy indication attended in Gynecological Surgery clinic of the Hospital Pedro I.

Sample

It will be obtained a non-consecutive probability sample offering to participate in the study to all women that is going to be submitted to total abdominal hysterectomy indication in the referral hospital from june 2015 to june 2016. Then these will be submitted to randomization process as explained later.

Calculation of the sample Size:

The calculation of sample size was performing using the online software in the public domain Openepi version 2.3.1 (Atlanta, GA). Were used as reference data found in clinical trial using gabapentin versus placebo (AJORI et al., 2011), in which it found an average of Visual Analog Scale score of 0.2 and a standard deviation of 0.8 for the group receiving gabapentin and average of 0.9 to 1.3 standard deviation for the group with placebo administration. For a power of 95% and a significance level of 5%, would require 124 patients (62 in each group) to highlight this difference. It is expected losses or post-randomization exclusion, was added to 20% of the total patients, resulting in 148.8 or approximately 150 patients (75 in each group).

Procedures for participants selection

Patients with total abdominal hysterectomy indication usually are hospitalized in the previous day in the hospital. They will be addressed by one of the researchers to apply a checklist with the criteria for inclusion and exclusion and, if eligible, will be invited to participate. The informed consent will be read aloud and those who agree to participate will then be randomized to one of the groups: amitriptyline or placebo.

Randomization Procedures

A list of random numbers will be previously prepared by a statistical oblivious to research in the public domain software Random Allocation Software version 2.0 (Ispaham, Iran), with 75 patients allocated to the amitriptyline group and 75 to the placebo group.

Boxes will be prepared to pack the tablets containing 25 mg of amitriptyline or placebo. Any amitryptyline as a placebo have been prepared by the hospital pharmacy with aspect (size, shape, weight and color) identical. Consecutively numbered boxes are packed in a 150 intended consecutively for each patient randomized. These boxes will be prepared by a pharmacist also oblivious to the research and researchers, and patients, will not be aware of its content, therefore ensuring it is the concealment of allocation.

Both tablets will be administered orally, with water being offered to patients in the period between six and twelve hours before the surgical procedure by the head nurse of the gynecology ward (blinded to the study), which should correspond to the nighttime for surgeries performed in the morning and the morning period for surgeries performed in the afternoon.

Data processing

The data collected should follow the following protocol for storage: should first occur data collection, followed by creation of a base number of patient follow-up with nine digits. The first six digits should refer to the day of collection in the day, month, year, each with two digits. The last three digits should be reserved to the sequence order in which the tests were performed. Thus, in the case of the first day the patient should be 001 if the second was 002 and so on. Eg patient number 070912005. It is known that was attended for the first time on 07/09/12 and that was the day the patient fifth part of the sample.

The data will be entered in a specific database created in the public domain Epi-Info 7.1.3 program and Medcalc version 13.2.2 or higher, at different times by two different people. After typing, the databases will be compared. Consistency tests and frequency distribution tables of the main variables will be obtained for any errors correction. In the case of finding inconsistencies or lack of information, the forms will be consulted. If doubt remains, will be made the consultation of the records.

At the end of typing, listings will be obtained again for the last correction and creating the final database, which will be submitted to cleaning tests and consistency of information, leading to the final database, which will be used for statistical analysis .

4.15.2 Data Analysis

Statistical analysis will be performed by researchers in the Epi-Info 7.1.3 and Medcalc version 13.2.2 or higher version available at the time, identifying the groups as A or B and breaking up the secrecy only after the results obtained and prepared the tables. Thus, only you know which group received amitriptyline or placebo at the end of the analysis.

The visual analogic scale can be recorded to binary mild / absent and moderate / severe pain pain, using cut-off points to be set later. It will also be analyzed as ordinal variable, using for comparison of the groups the nonparametric Mann-Whitney test. The same procedure is used to evaluate the satisfaction and depression, thereby obtaining categorical variables.

Categorical variables are compared in contingency tables using the chi-square tests of association and Fisher's exact test where appropriate. It will calculate the risk ratio (RR) as a relative measure of risk, determining the 95% confidence interval. The numbers needed to treat and get a benefit and number needed to treat and get a harm will still be calculated and their respective confidence intervals at 95%.

At every stage of the analysis will be adopted the significance level of 5%.

Ethics aspects

This study meets the requirements of the "Declaration of Helsinki" for research on human subjects, and Resolution 466/2012 of the National Health Council (BRAZIL MINISTRY OF HEALTH, 2012).

All participants will be informed about the research objectives and with free will to their participation or not. The participants will be informed about possible side effects and at the same time the possible beneficial effects of amitriptyline, being informed that they will not be aware will be using this drug or placebo. Patients should also be aware that any damage suffered can and preferably should be reported immediately to one of the evaluators. Example: adverse reaction to amitriptyline not provided in the package leaflet.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for total abdominal hysterectomy for benign conditions (e.g. hemorrhagic and / or uterine fibroid disorder);
* Age between 18 and 60;

Exclusion Criteria:

* Endometriosis;
* Abnormal cervicovaginal smears;
* Uterine prolapse;
* Patients with a history of intolerance to opioids or narcotics;
* Patients with contraindications to the use of amitriptyline (e.g., ischemic heart disease, glaucoma)
* addicted to alcohol or drugs;
* Use of analgesics in the 24 hours prior to the possible administration of amitriptyline;
* Failure to provide informed consent;
* Different anesthesia from spinal anesthesia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of amitryptyline in the prevention of post-operative pain in women undergoing total abdominal hysterectomy, twenty-four hours after surgery | Twenty-four hours after surgery
  The postoperative pain will be measured twenty-four hours after surgery, using the visual pain scale (0 - no pain to 10 - very hard pain)

SECONDARY OUTCOMES:
Intensity of acute postoperative pain six hours after the procedure | Six hours after the procedure
  It will be measured using the visual pain scale (0 - no pain to 10 - very hard pain)
Intensity of acute postoperative pain twelve hours after the procedure | Twelve hours after the procedure
  It will be measured using the visual pain scale (0 - no pain to 10 - very hard pain)
Intensity of acute postoperative pain twenty-four hours after the procedure | Twenty-four hours after the procedure
  It will be measured using the visual pain scale (0 - no pain to 10 - very hard pain)
Intensity of acute postoperative pain forty-eight hours after the procedure | forty-eight hours after the procedure
  It will be measured using the visual pain scale (0 - no pain to 10 - very hard pain)
Records of rescue analgesia | From the end of the procedure until 48 hours after that
  Use of rescue analgesia with the infusion of morphine - It will be checked using the patient records at the hospital
Compare surgical time (duration, in minutes) and frequency of intraoperative and postoperative complications | From the end of the procedure until sixty days after that.
  Relationship between surgical time (duration) and complications occurrence
Frequency of adverse effects | From the end of the procedure until 48 hours after that
  Onset of adverse effects like migraine, sickness, numbness, vomiting, itching, etc
Length of hospitalization | participants will be followed for the duration of hospital saty, an expected average of 48 hours.
  Time between admission and releasing, in hours
Effectiveness of amitryptyline in the prevention of post-operative pain in women undergoing total abdominal hysterectomy, six hours after surgery | Six hours after surgery.
  The postoperative pain will be measured after six hours after surgery, using the visual pain scale (0 - no pain to 10 - very hard pain)
Effectiveness of amitryptyline in the prevention of post-operative pain in women undergoing total abdominal hysterectomy, twelve hours after surgery | Twelve hours after surgery
  The postoperative pain will be measured after six hours after surgery, using the visual pain scale (0 - no pain to 10 - very hard pain)
Effectiveness of amitryptyline in the prevention of post-operative pain in women undergoing total abdominal hysterectomy, forty-eight hours after surgery | Forty-eight hours after surgery
  The postoperative pain will be measured forty-eight hours after surgery, using the visual pain scale (0 - no pain to 10 - very hard pain)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme V Mascena, PhD, Study Chair — FCM-CG
Locations (1):
- FCM CG - Faculdade de Ciências Médicas de Campina Grande, Campina Grande, Paraíba, Brazil

REFERENCES:
- [Background] Arsenault A, Sawynok J. Perisurgical amitriptyline produces a preventive effect on afferent hypersensitivity following spared nerve injury. Pain. 2009 Dec;146(3):308-314. doi: 10.1016/j.pain.2009.08.003. Epub 2009 Sep 11. PMID 19748184
- [Background] Brandsborg B. Pain following hysterectomy: epidemiological and clinical aspects. Dan Med J. 2012 Jan;59(1):B4374. PMID 22239844
- [Background] Buvanendran A, Kroin JS, Della Valle CJ, Kari M, Moric M, Tuman KJ. Perioperative oral pregabalin reduces chronic pain after total knee arthroplasty: a prospective, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):199-207. doi: 10.1213/ANE.0b013e3181c4273a. Epub 2009 Nov 12. PMID 19910619
- [Background] Clarke-Pearson DL, Geller EJ. Complications of hysterectomy. Obstet Gynecol. 2013 Mar;121(3):654-673. doi: 10.1097/AOG.0b013e3182841594. PMID 23635631
- [Background] Goodwin SA. A review of preemptive analgesia. J Perianesth Nurs. 1998 Apr;13(2):109-14. doi: 10.1016/s1089-9472(98)80095-6. PMID 9592452
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Moiniche S, Kehlet H, Dahl JB. A qualitative and quantitative systematic review of preemptive analgesia for postoperative pain relief: the role of timing of analgesia. Anesthesiology. 2002 Mar;96(3):725-41. doi: 10.1097/00000542-200203000-00032. No abstract available. PMID 11873051
- [Result] Ajori L, Nazari L, Mazloomfard MM, Amiri Z. Effects of gabapentin on postoperative pain, nausea and vomiting after abdominal hysterectomy: a double blind randomized clinical trial. Arch Gynecol Obstet. 2012 Mar;285(3):677-82. doi: 10.1007/s00404-011-2023-6. Epub 2011 Aug 5. PMID 21818576